CLINICAL TRIAL: NCT02113813
Title: An Open-label, Phase 1 Dose Escalation Study of Oral ASP8273 in Subjects With Non-Small-Cell Lung Cancer (NSCLC) Who Have Epidermal Growth Factor Receptor (EGFR) Mutations
Brief Title: A Dose Escalation Study of ASP8273 in Subjects With Non-Small-Cell Lung Cancer (NSCLC) Who Have Epidermal Growth Factor Receptor (EGFR) Mutations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8273-CL-0102
Record Dates: First submitted 2014-04-04; First posted 2014-04-15 (Estimated); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Non-Small-Cell Lung Cancer (NSCLC); Epidermal Growth Factor Receptor Mutations
Keywords: irreversible EGFR inhibitor; Non-Small-Cell Lung Cancer; Midazolam; T790M resistance mutation; EGFR; NSCLC; naquotinib; Epidermal Growth Factor Receptor mutations; ASP8273
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — naquotinib; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- ASP8273 Dose Escalation cohort (part 1) (Experimental): oral
  Interventions: Drug: naquotinib
- ASP8273 Response Expansion cohort (part 1) (Experimental): oral
  Interventions: Drug: naquotinib
- ASP8273 and Midazolam RP2D Expansion cohort (part 2) (Experimental): oral
  Interventions: Drug: naquotinib; Drug: midazolam
- Food Effect Fasted cohort (part 2) (Experimental): oral
  Interventions: Drug: naquotinib
- Food Effect Fed cohort (part 2) (Experimental): oral
  Interventions: Drug: naquotinib
- Exon 20 Cohort (part 2) (Experimental): oral
  Interventions: Drug: naquotinib

INTERVENTIONS:
Drug: naquotinib — oral
  Other Names: ASP8273
Drug: midazolam — oral
  Arms: ASP8273 and Midazolam RP2D Expansion cohort (part 2)

SUMMARY:
The purpose of this study is to assess the safety and tolerability of ASP8273 and to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D). This study will also determine the pharmacokinetics (PK) of ASP8273, evaluate the potential inhibition of CYP3A4 by ASP8273 and the antitumor activity of ASP8273 as well as determine the effect of food on the bioavailability of ASP8273.

DETAILED DESCRIPTION:
This study is composed of 2 parts: part 1 is the dose escalation phase and part 2 is the recommended Phase 2 dose (RP2D) phase, Food Effect (FE) cohort and Exon 20 cohort.

ELIGIBILITY:
Inclusion Criteria:

* Non-child bearing potential or able to follow birth control requirements
* Eastern Cooperative Oncology Group (ECOG) ≤ 1
* Life expectancy ≥ 12 weeks
* Laboratory criteria as:

  * Neutrophil count ≥ 1,500/mm3
  * Platelet count ≥ 7.5 x 104 /mm3
  * Hemoglobin ≥ 9.0 g/dL
  * Lymphocyte count ≥ 500/mm3
  * Serum creatinine < 1.5 x institutional Upper Limit of Normal (ULN) or an estimated glomerular filtration rate (eGFR) of > 50 ml/min as calculated by the Modification of Diet in Renal Disease (MDRD) equation
  * Total bilirubin < 1.5 x ULN (except for subjects with documented Gilbert's syndrome)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3.0 x ULN
* Dose escalation subjects: Epidermal Growth Factor Receptor (EGFR) activating mutation by local testing: exon 18 G719X, exon 19 deletion, exon 21 L861Q, exon 21 L858R or exon 20 insertion; and received prior treatment with EGFR Tyrosine Kinase Inhibitor (TKI)
* Response expansion/RP2D expansion/ FE Cohort subjects: disease progression on or was intolerant to prior EGFR TKI; activating mutation as above AND T790M mutation; tumor sample subsequent to EGFR TKI is available for central testing; at least one measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1

Inclusion Criteria for Exon 20 cohort:

* Subject on any line of treatment and has an EGFR exon 20 insertion mutation on examination of an NSCLC tissue or cellular specimen. Local testing may determine eligibility and a tumor sample should also be sent for central testing.
* Subjects must have at least 1 measurable lesion based on RECIST version 1.1.

Exclusion Criteria:

* Any ongoing toxicity ≥ Grade 2 attributable to prior Non-Small-Cell Lung Cancer (NSCLC) treatment
* Prior EGFR inhibitor within 6 days; received prior treatment with any other agent with antitumor activity chemotherapy, radiotherapy, or immunotherapy within 14 days; any investigational therapy within 28 days or 5 half-lives, whichever is shorter; blood transfusion or hemopoietic factor within 14 days; major surgery within 14 days; any strong CYP3A4 inhibitors within 7 days
* Positive hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) or Human Immunodeficiency Virus (HIV)
* Symptomatic Central Nervous System (CNS) metastasis
* Active infection requiring systemic therapy within 14 days
* Severe or uncontrolled systemic diseases including uncontrolled hypertension
* History of or active interstitial lung disease
* Screening QTcF >450 msec or current medication known to prolong QT
* ≥ Grade 2 cardiac arrhythmia or uncontrolled atrial fib of any grade; Class 3 or 4 New York Heart Association congestive heart failure; history of severe/unstable angina, myocardial infarction or cerebrovascular accident within 6 months
* History of gastrointestinal ulcer or bleeding within 3 months; any digestive tract dysfunction
* Concurrent corneal disorder or ophthalmologic condition making subject unsuitable
* RP2D cohort subjects: contraindications to midazolam, any other midazolam within 7 days, or any medications or supplements known to be strong CYP3A inhibitors within 7 days or inducers within 12 days
* Any other malignancy requiring treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2014-04-09 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by Dose Limiting Toxicities (DLTs) | up to 18 months
  A DLT is defined as any pre-determined toxicity that is related to study drug per the investigator and which occurs during Cycle 0 and Cycle 1 using NCI CTCAE v4.03.
Safety and tolerability as assessed by adverse events (AEs) | up to 18 months
  An AE is defined as any untoward medical occurrence in a subject administered a study drug or has undergone study procedures and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Safety and tolerability as assessed by laboratory tests | up to 18 months
  Laboratory tests to be conducted are hematology, biochemistry, urinalysis, coagulation profile, lipid panel and lymphocyte subpopulation.
Safety and tolerability as assessed by vital signs | up to 18 months
  Vital signs to be measured includes blood pressure, pulse rate and temperature.
Safety and tolerability as assessed by 12-lead electrocardiograms (ECGs) | up to 18 months

SECONDARY OUTCOMES:
Composite of pharmacokinetics of ASP8273 concentration and its metabolites (plasma): Cmax, tmax, AUClast, AUCinf, t1/2, CL/F, and Vz/F | Cycle 0: Dose Escalation Days 1-2, FE Days 1-6; Cycle 1: Dose Escalation/Response Expansion/RP2D/FE Days 1,8,15, RP2D Day 21, Exon 20 Days 8,15; Cycle 2 & 3: Dose Escalation/Response Expansion/RP2D Days 1,2, FE Day 1; Exon 20 days 1, 2 & Cycle 3
  Maximum concentration (Cmax), the time after dosing when Cmax occurs (tmax), area under the concentration - time curve from time 0 up to the last quantifiable concentration (AUClast), area under the concentration - time curve from time 0 extrapolated to infinity (AUCinf), apparent terminal elimination half-life (t1/2), apparent oral systemic clearance (CL/F), Apparent volume of distribution (Vz/F)
Composite of pharmacokinetics of midazolam concentration and its metabolites (plasma): Cmax, tmax, AUClast, AUCinf, t1/2, CL/F, and Vz/F | Day -1 and Day 1 of cycle 1; Day 1 and Day 2 of cycle 2
Best overall response rate | Up to 18 months
  Defined as proportion of subjects whose best overall response is Complete Response (CR) or Partial Response (PR) among all analyzed subjects.
Disease control rate | Up to 18 months
  Defined as the proportion of subjects whose best overall response is rated as CR, PR or Stable Disease (SD) among all analyzed subjects.
Progression free survival | Up to 18 months
  Defined as the time from the start of the study treatment until death from any cause or radiographic disease progression assessed according to RECIST 1.1, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (12):
- United States (12):
  - Site US10010, Washington D.C., District of Columbia
  - Site US10006, Baltimore, Maryland
  - Site US10012, Boston, Massachusetts
  - Site US10001, Boston, Massachusetts
  - Site US10011, Boston, Massachusetts
  - Site US10008, New York, New York
  - Site US10004, Chapel Hill, North Carolina
  - Site US10005, Cleveland, Ohio
  - Site US10009, Philadelphia, Pennsylvania
  - Site US10002, Nashville, Tennessee
  - Site US10003, Fairfax, Virginia
  - Site US10007, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=342